CLINICAL TRIAL: NCT00361036
Title: Feasibility Evaluation of the Embolic Agent BeadBlock™ in the Treatment of Uterine Fibroids With Uterine Artery Embolization With Comparison of Study Endpoints to Embosphere®
Brief Title: Comparison Study in the Treatment of Uterine Fibroids Uterine Fibroid Embolization Using BeadBlock™ Embolic Agent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Worthington-Kirsch, Robert L., M.D. (Individual)
Collaborators: Terumo Medical Corporation (Industry); Biocompatibles UK Ltd (Industry)
Responsible Party: Robert Worthington-Kirsch MD, Image Guided Surgery associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G060030
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Leiomyoma; Leiomyomatosis; Uterine Neoplasms
Keywords: Leiomyoma; Leiomyomatosis; Uterine Neoplasms; BeadBlock; Embsophere; Embolization; Uterine fibroid embolization
MeSH Terms: conditions — Leiomyoma; Leiomyomatosis; Uterine Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): BeadBlock treatment arm
  Interventions: Device: Uterine fibroid embolization BeadBlock™
- 2 (Active Comparator): Embospheres control arm
  Interventions: Device: Uterine fibroid embolization Embosphere®

INTERVENTIONS:
Device: Uterine fibroid embolization BeadBlock™ — Intervention with BeadBlock Microspehere
  Arms: 1
Device: Uterine fibroid embolization Embosphere® — Embosphere - control arm
  Arms: 2

SUMMARY:
A double arm (non-inferiority) 44 patient study to assess the performance of BeadBlock™ in the treatment of uterine fibroids by embolization with respect to clinical & imaging outcome with comparison of primary safety endpoints to Embosphere.

DETAILED DESCRIPTION:
The purpose of the study is to conduct a comparison between BeadBlock™ and Embosphere in uterine fibroid embolization. Baseline and follow-up MR Imaging data will be made with respect to changes in fibroid and uterus perfusion and fibroid and uterine volume. This is a 12 months study (12 month follow up for all enrollees). The primary end-point will be the degree of fibroid devascularization as seen at contrast-enhanced MRI performed 3 months (+/- 15 days) after UAE procedure. In addition we will assess symptom reduction in patients that have undergone uterine fibroid embolization with Bead Block™ and Embosphere®.

Primary Objective 1. To assess the change in fibroid devascularization as seen at contrast-enhanced MRI performed after UAE and at three (3) months (+/- 15 days) following the UAE, and compare the changes between BeadBlock™ and Embosphere.

Secondary Objective

1. To assess the change in fibroid devascularization as seen at contrast-enhanced MRI performed several days after UAE and 6 months (+/- 15 days) following the UAE, and compare the changes between BeadBlock™ and Embosphere.

Tertiary Objective

1. To assess the change in uterine volume as seen at contrast-enhanced MRI performed several days after UAE, 3 months (+/- 15 days) and 6 months (+/- 15 days) following the UAE, and compare the changes between BeadBlock™ and Embosphere.
2. To assess the change from baseline in symptom severity (UFS-QOL)at 3, 6 and 12 months (+/- 15 days) follow-up, as measured by the subscale of the UFS questionnaire, and compare the changes between BeadBlock™ and Embosphere.

ELIGIBILITY:
Inclusion Criteria:

1. Patient chooses to participate and has signed informed consent
2. Age between 30 and 50 years old
3. Symptoms caused by uterine fibroids, such as heavy bleeding (menorrhagia) and/or bulk-related complaints such as urinary frequency, constipation or pelvic pain.
4. Patient has fibroids confirmed by MRI
5. Patient has normal kidney function.
6. Patient is willing and able to undergo follow-up imaging at 3 and 6 months post UFE.

Exclusion Criteria:

1. Patients who are pregnant or plan to become pregnant within the study period, or desire future fertility.
2. Patients with a history of gynecologic malignancy
3. Patients with known endometrial hyperplasia
4. Patients with adenomyosis
5. Patients with pelvic inflammatory disease
6. Patients with Uteri < 250 ml (cm) calculated volume or > 24 weeks
7. Patients with pedunculated subserosal fibroids with a narrow attachment (<50% diameter of the fibroid) to the uterus.
8. Patients with pelvic pain as dominant syndrome
9. Known allergy to contrast media that cannot be adequately pre-medicated.
10. Patients not suitable for arterial access.
11. Previous uterine artery embolization attempts.
12. History of pelvic irradiation.
13. Patients on GnRH Therapy within 3-6 months prior to the study enrollment.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in fibroid devascularization as seen at contrast enhanced MRI performed several days after UAE and 3 months following the UAE between BeadBlock™ and Embosphere | 12 months

SECONDARY OUTCOMES:
Mean difference of change in fibroid devascularization CEMRI performed several days after UAE and 6 months following the UAE between BeadBlock™ and Embosphere. | 12 months
assess the change from baseline in symptom severity (UFS-QOL)at 3, 6 and 12 months (+/- 15 days) follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Worthington-Kirsch, MD, Principal Investigator — Image Guided Surgery Associates
Locations (2):
- United States (2):
  - Albany Medical Center, Albany, New York
  - Image Guided Surgery Associates, Pottstown, Pennsylvania

REFERENCES:
- [Derived] Worthington-Kirsch RL, Siskin GP, Hegener P, Chesnick R. Comparison of the efficacy of the embolic agents acrylamido polyvinyl alcohol microspheres and tris-acryl gelatin microspheres for uterine artery embolization for leiomyomas: a prospective randomized controlled trial. Cardiovasc Intervent Radiol. 2011 Jun;34(3):493-501. doi: 10.1007/s00270-010-0049-y. Epub 2010 Dec 3. PMID 21127866
- See also: Management of Uterine fibroids Summary report — http://www.ahrq.gov/clinic/epcsums/utersumm.htm
- See also: Emmy Trial: Uterine Artery Embolization (UAE) Versus Hysterectomy for Uterine Fibroids — http://www.clinicaltrials.gov/ct/show/NCT00100191
- See also: Uterine artery embolization versus hysterectomy in the treatment of symptomatic uterine fibroids (EMMY trial): peri- and postprocedural results from a randomized controlled trial — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=PubMed&dopt=Abstract&list_uids=16260201